CLINICAL TRIAL: NCT00998816
Title: A Multicenter Prospective Randomized Double-blind Placebo Controlled Trial Assessing the Effect of Perioperative Pregabalin on the Incidence of Chronic Post Thoracotomy Pain Syndrome
Brief Title: The Effect of Perioperative Pregabalin on the Incidence of Chronic Post-thoracotomy Pain Syndrome
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No funding
Sponsor: Queen's University (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Jorge Zamora, Associate Professor, MD, FRCPC, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ANAE 153-09
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Pain
Keywords: thoracotomy; chronic; pain; pregabalin; Lyrica
MeSH Terms: conditions — Chronic Pain; Bronchiolitis Obliterans Syndrome; Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo capsules (Placebo Comparator): one placebo capsule will be administered 1 hour before lateral thoracotomy, 12 hours following the thoracotomy and then every 12h BID for 10 days following lateral thoracotomy.
  Interventions: Drug: Pregabalin
- pregabalin capsules (Active Comparator): Pregabalin capsules (150mg) will be administered one hour before lateral thoracotomy, 12 hours following the thoracotomy and then every 12 hours (BID) for 10 days following lateral thoracotomy.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — pregabalin capsules (150mg,oral) will be administered 1 hour before lateral thoracotomy, 12 hours after the thoracotomy and then 12 h BID for 10 additional days.
  Other Names: Lyrica

SUMMARY:
Pregabalin, administered prior to and following lateral thoracotomy surgery will reduce the likelihood of chronic post-thoracotomy pain syndrome (CPTPS).

DETAILED DESCRIPTION:
A total of 200 patients scheduled for lateral thoracotomy will be randomly assigned to receive either placebo or 150 mg pregabalin (Lyrica)1 hour prior to surgery, 12 hr after surgery and then every 12 hr for an additional 10 days. While in the hospital, patients will be assessed for pain intensity, satisfaction and side effects. Patients will be re-assessed at 2, 4 and 6 months following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective open thoracotomy for primary thoracic surgery, understanding and provision of written informed consent, ASA class I II or III

Exclusion Criteria:

* Inability ot adhere to study protocol:

  * intolerance or hypersensitivity to any agents to be used in the study, contraindication to thoracic epidural placement
  * inability to respond to the study questionnaire
  * renal insufficiency(serum creatinine > 1.5 upper limit of normal)
  * Body Mass index > 40
  * planned post-operative ventilation.
* Confounding procedural factors which might affect validity of data:

  * previous ipsilateral thoracotomy
  * surgery for tumor extending into the chest wall
  * rest pain in proposed surgical area pre-operatively
  * chest tube in situ at time of surgery
  * requirement for second thoracotomy or re-occurrence of disease after surgery *isolated pleuroscopy or pleurodesis procedures.
* Potential interaction with study medications and patient's current medications:

  * current alcohol or other substance abuse
  * chronic steroid use
  * pre-existing chronic pain requiring chronic analgesic use
  * history of seizure disorder requiring treatment with an anticonvulsant
  * current therapy with thiazolidinedione class oral hypoglycemic agents (eg, Actos, Avandia or Avandamet)
  * history of congestive heart failure
  * major psychiatric disorder
  * any contraindication to use of NSAIDs.
* Insufficient safety data in the patient population:

  * patients requiring preoperative assistance or assistive device for ambulation, pregnant or breastfeeding
  * weight <50 Kg
  * dizziness while inpatient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic post thoracotomy pain syndrome | 6 months following surgery

SECONDARY OUTCOMES:
During hospital stay: pain intensity, PEF and FEV1, patient satisfaction, medication side effects. At 2, 4, and 6 months: pain intensity, pain quality (neuropathic versus other), quality of life, pain interference with daily function | During hospital stay and at 2, 4, and 6 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Zamora, MD, Principal Investigator — Queen's University/ Kingston General Hospital
Locations (1):
- Dr. Jorge E Zamora, Kingston, Ontario, Canada